CLINICAL TRIAL: NCT00005917
Title: Investigations Into Chediak-Higashi Syndrome and Related Disorders
Brief Title: Study of Chediak-Higashi Syndrome
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000153; 00-HG-0153
Record Dates: First submitted 2000-06-16; First posted 2000-06-19 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-07-08

CONDITIONS: Chediak-Higashi Syndrome
Keywords: Albinism; Giant Granules; Infection; Melanosomes; Platelet Storage Pool Defect; Natural History
MeSH Terms: conditions — Chediak-Higashi Syndrome; Albinism; Infections; Platelet Storage Pool Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chediak-Higashi Syndrome: Confirmed or suspected patients with Chediak-Higashi Syndrome.

SUMMARY:
Chediak-Higashi syndrome (CHS) is a rare autosomal recessive disorder characterized in its classical form by oculocutaneous albinism, a bleeding diathesis, recurrent infection due to abnormal neutrophil and natural killer cell function, and eventual progression to a lymphohistiocytic infiltration known as the accelerated phase . Death often occurs within the first decade as a result of infection or the development of the accelerated phase; bone marrow transplantation is curative except for the late occurrence of neurological deterioration. The basic defect is unknown, although it probably involves abnormal fusion or trafficking of intracellular vesicles. Patients with classical CHS have their disease due to mutations in the LYST gene, but mildly affected individuals have been reported whose genetic defect has not been defined. It is likely that these variants of CHS have abnormalities in proteins involved in the pathways responsible for vesicle fusion. Since the full clinical spectrum of CHS and its variants has not been characterized, and the underlying defects remain enigmatic, we plan to evaluate this group of patients clinically, biochemically, and molecularly, and perform cell biological studies on their fibroblasts, melanocytes, and transformed lymphoblasts. Routine admissions will be 5 days and may occur every two years, or required by changes in clinical symptomatology....

DETAILED DESCRIPTION:
Chediak-Higashi syndrome (CHS) is a rare autosomal recessive disorder characterized in its classical form by oculocutaneous albinism, a bleeding diathesis, recurrent infection due to abnormal neutrophil and natural killer cell function, and often progression to a lymphohistiocytic infiltration known as the accelerated phase . Death generally occurs within the first decade as a result of infection or the development of the accelerated phase; bone marrow transplantation is curative except for the late occurrence of neurological deterioration. However, our research has identified mildly affected individuals who present primarily with a neurological phenotype characterized by central and peripheral nervous system involvement. In addition, classical cases treated with bone marrow transplant (BMT) and surviving into adulthood usually develop neurological symptoms adding relevance to the study of pathophysiology of this disease outside of the hematological and immune systems. The only gene known to be associated with CHS is LYST; however, there are some patients with CHS in whom mutations have not been found, suggesting locus heterogeneity. A genotype-phenotype correlation had begun to emerge, but recent reports noted exceptions to this correlation. The basic defect is unknown, although it probably involves abnormal fusion or trafficking of intracellular vesicles. With regards to neurologic involvement, LYST likely also plays a role in neuronal axonal transport and neurotransmitter pools. We plan to evaluate individuals with CHS clinically, biochemically, and molecularly, and perform cell biological studies on their fibroblasts, melanocytes, and transformed lymphoblasts. Routine admissions may be 3-5 days and may occur every one to two years, or as required by changes in clinical symptomatology.

ELIGIBILITY:
* ELIGIBILITY:

Patients will be between the age of 1 month and 70 years. All patients entering this study will have some degree of oculocutaneous albinism plus either a bleeding diathesis or a history of excessive infections in childhood. Objective evidence of a platelet storage pool deficiency (e.g., an abnormal secondary aggregation response or absent platelet dense bodies) or of a lysosomal fusion abnormality (e.g., giant cytoplasmic granules in leucocytes) will not be required.

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients entering this study will have clinical features suggestive of CHS. Objective evidence of a platelet storage pool deficiency (e.g., an abnormal secondary aggregation response or absent platelet dense bodies) or of a lysosomal fusion abnormality (e.g., giant cytoplasmic granules in leucocytes) will not be required.@@@
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2002-09-10 (Actual)

PRIMARY OUTCOMES:
Delineate the clinical and laboratory findings of CHS and its variants. | 4-5 days every 1-2 years
  Delineate the clinical and laboratory findings of CHS and its variants.

SECONDARY OUTCOMES:
Mutation analysis of the LYST gene will be performed, to further delineate genotype/phenotype correlations and or locus heterogeneity. | 4-5 days every 1-2 years
  Mutation analysis of the LYST gene will be performed, to further delineate genotype/phenotype correlations and or locus heterogeneity.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Introne, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This data will be deidentified.
Supporting Information: Study Protocol
Time Frame: While the study is open.
Access Criteria: All data sharing will be approved by the NHGRI Tech Transfer Office.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2000-HG-0153.html